CLINICAL TRIAL: NCT01469104
Title: Metabolic Response to 3-day Fast Versus Carbohydrate-free Diet in Type 2 Diabetes
Acronym: CHO-free diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Frank Q. Nuttall, MD, PhD, Chief, Endocrinology, Metabolism & Nutrition Section, Professor of Medicine, Minneapolis Veterans Affairs Medical Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 4177
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2011-11-10 (Estimated); Status verified 2011-11

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 3 day fast (Placebo Comparator): After receiving a standard diet on day 1, subject will fast on days 2, 3, and 4. Water and calorie-fee beverages will be allowed during this 72 hour period.
  Interventions: Other: 3 day fast
- CHO-free diet (Active Comparator): After receiving a standard diet on day 1, a carbohydrate-free diet will be provided on days 2, 3, and 4.
  Interventions: Other: 3 day CHO-free diet

INTERVENTIONS:
Other: 3 day fast — Subjects will fast for 72 hours
  Other Names: 3-Day Fast
  Arms: 3 day fast
Other: 3 day CHO-free diet — Subjects will receive a carbohydrate-free diet for 72 hours
  Other Names: Carbohydrate-free diet
  Arms: CHO-free diet

SUMMARY:
The investigators hypothesis is that a carbohydrate-free diet, ingested for 3 days, results in a change in blood glucose that is similar to the change observed after 3 days of fasting.

DETAILED DESCRIPTION:
In addition to plasma glucose concentrations, other hormones and metabolites known to be affected by fasting will be measured. These include insulin and glucagon, which are hormones that have an important role in regulating fuel use in the body.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* C-peptide > 1.5 ng/ml

Exclusion Criteria:

* Body mass index > 40
* hematological abnormalities
* liver disease
* kidney disease
* congestive heart failure
* life threatening malignancies

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-08; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Change in plasma glucose concentration | 24 hour profile:before and after meals, or traditional meal times

SECONDARY OUTCOMES:
Change in serum insulin concentrations | 24 hour profiles: before and after meals or traditional meal times

CONTACTS AND LOCATIONS:
Overall Officials: Frank Q. Nuttall, M.D., Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center; Mary C. Gannon, Ph.D., Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Nuttall FQ, Almokayyad RM, Gannon MC. The ghrelin and leptin responses to short-term starvation vs a carbohydrate-free diet in men with type 2 diabetes; a controlled, cross-over design study. Nutr Metab (Lond). 2016 Jul 22;13:47. doi: 10.1186/s12986-016-0106-x. eCollection 2016. PMID 27453716
- [Derived] Nuttall FQ, Almokayyad RM, Gannon MC. Comparison of a carbohydrate-free diet vs. fasting on plasma glucose, insulin and glucagon in type 2 diabetes. Metabolism. 2015 Feb;64(2):253-62. doi: 10.1016/j.metabol.2014.10.004. Epub 2014 Oct 8. PMID 25458830